CLINICAL TRIAL: NCT02501616
Title: Effect of Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor on Systemic and Renal Endothelial Function in Patients With Type 2 Diabetes Mellitus Without History of Coronary Artery Disease (SOCCER Trial)
Brief Title: Effect of Dapagliflozine on Systemic and Renal Endothelial Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Min Kyong Moon, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BRMH 26-2014-148
Record Dates: First submitted 2015-07-12; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Endothelial Function; Type 2 Diabetes
Keywords: SGLT2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; dapagliflozin

ARMS (2):
- Metformin first (Active Comparator): Metformin first 8 wks --> Dapagliflozin 8wks.
  Metformin for initial 8 weeks. During that period, metformin can be titrated upto 2000 mg/day. After 1 weeks of washout period, 8 weeks' dapagliflozin is followed. During that period, dose of dapagliflozin is maintained 10mg/day.
  Interventions: Drug: Metformin; Drug: Dapagliflozin
- Dapagliflozin first (Active Comparator): Dapagliflozin first 8 wks --> Metformin 8wks.
  Dapagliflozin for initial 8 weeks. After 1 weeks of washout period, 8 weeks' metformin is followed.
  Interventions: Drug: Metformin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Metformin
Drug: Dapagliflozin
  Other Names: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor

SUMMARY:
This is a phase 4, single center, randomized, open-labeled, cross-over design study. The primary objective of the study is to compare effect of dapagliflozine and metformin on endothelial function.

Subjects are randomized to initial metformin or initial dapagliflozin group and maintained initial treatment for 8 weeks. During that period, dose of dapagliflozin is maintained 10mg/day and metformin can be titrated upto 2000 mg/day. After 1 weeks of washout period, 8 weeks' cross-over is followed.

ELIGIBILITY:
Inclusion Criteria:

1. Present with type 2 diabetes based on the disease diagnostic criteria as described by the World Health Organization (WHO)
2. Treated with diet and exercise alone for recent 3 months
3. Aged 20-80 years
4. HbA1c 7~9%
5. This inclusion criterion applies to females of childbearing potential (not surgically sterilized and between menarche and 1-year postmenopause) only.

   * Are not breastfeeding.
   * Test negative for pregnancy at the time of screening based on a blood serum pregnancy test.
   * Intend not to become pregnant during the study.

Exclusion Criteria:

1. Previous history of IHD or brain infarct
2. Having typical anginal pain or atypical chest pain with dyspnea
3. Modification of Diet in Renal Disease (MDRD) estimated GFR≥60 mL/min

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Reactive hyperemic index to measure endothelial function | 8 weeks
  endothelial function

SECONDARY OUTCOMES:
N-acetyl-β-D-glucosaminidase as a measure of renal tubular injury | 8 week
  renal tubular injury
Urine albumin excretion ratio | 8 week
  Urine albumin excretion
Urine β2 microglobulin | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyong Moon, MD PhD, Principal Investigator — Boramae medical center, 20 Boramae-ro 5-gil,Dongjak-Gu,Seoul 156-707, Korea
Locations (1):
- Boramae medical center, Seoul, South Korea